CLINICAL TRIAL: NCT01603706
Title: Radial Strain Imaging-Guided Lead Placement for Improving Response to Cardiac Resynchronization Therapy in Patients With Ischemic Cardiomyopathy: A Randomized Clinical Trial
Brief Title: Radial Strain ECHO-Guided Implantation of Cardiac Resynchronization Therapy
Acronym: RAISE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Rabin Medical Center (Other); Rambam Health Care Campus (Other); Kaplan Medical Center (Other); Soroka University Medical Center (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Prof. Michael Glikson, Prof. Michael Glikson, MD., Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-12-9349-MG-CTIL
Record Dates: First submitted 2012-05-14; First posted 2012-05-22 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Cardiomyopathy
Keywords: Heart failure; Cardiac Resynchronization Therapy; CRT; Radial strain echocardiography; Ischemic cardiomyopathy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Echo guided implantation group (Active Comparator): Echo guided implantation group Patients undergoing speckle tracking based LV lead implantation.
  Interventions: Procedure: Echo guided implantation group
- Conventional implantation group (No Intervention): Patients undergoing conventional LV lead implantation

INTERVENTIONS:
Procedure: Echo guided implantation group — Lead placement according echo strain imaging result
  Arms: Echo guided implantation group

SUMMARY:
The purpose of this study is to evaluate the use of radial strain imaging using speckle tracking analysis to predict the response to CRT in patients with ischemic cardiomyopathy (ICMP) with NYHA functional class 2-4 heart failure and a standard guideline-based CRT indication. Thus assessing the value of lead localization determined by radial strain imaging in a prospective, randomized manner.

DETAILED DESCRIPTION:
In this study we propose to evaluate the utility of radial strain imaging using speckle tracking to predict the response to CRT in patients with ischemic cardiomyopathy (ICMP) with NYHA functional class 2-4 heart failure and a standard guideline-based CRT indication, and to determine the value of lead localization determined by radial strain imaging in a prospective, randomized manner. We will compare two randomized groups of CRT recipients implanted with CRT-D systems. In the control group, implantation will be performed in the usual manner and the lead will be placed at the discretion of the implanting physician, preferably at posterolateral LV sites . In the study group, leads will be placed in areas of latest contraction that lack significant scar, as determined by speckle tracking imaging. The primary outcome measure for comparison between the 2 groups will be echocardiographic response (as assessed by percent reduction in left ventricular end systolic volumes) at 6 months post-implantation. In addition, clinical response parameters will also be measured as secondary end points.

We hypothesize that 1) patients showing greater dyssynchrony and/or discoordination index with speckle tracking will derive a significantly greater response to cardiac resynchronization therapy; and 2) patients allocated to the image-guided LV lead placement group will derive a significantly greater response to CRT than patients in the non- guided implantation (control) group.

If radial strain imaging proves useful for improving the CRT response rate and identification of patients likely to respond, it will have important clinical and economic implications by improving individual outcomes and more effective utilization of constrained health care resources. Furthermore, if echo-guided lead implantation proves to be effective in reducing the relatively large non-response rate to cardiac resynchronization therapy, it will likely result in increased device utilization among eligible heart failure patients.

Specific Aims Aim #1: To show that in patients with ischemic cardiomyopathy, implantation of a CRT LV lead guided by radial strain imaging results in a significantly greater echocardiographic and clinical response to cardiac resynchronization therapy compared with conventional implantation techniques.

Aim #2: To show that speckle tracking strain data can be used to identify the degree of echocardiographic response to CRT, using both dyssynchrony (time to peak strain ) and discoordination indices.

Aim #3:

The Paieon substudy will comprise 40 patients enrolled at 3 centers, for whom additional information mechanical dyssynchrony, using the Paieon CardioGuide motion map, will be collected during device implantation as detailed below The primary aim of the study is to relate data of mechanical dyssynchrony obtained from angiography through the Paieon CardioGuide motion map to dyssynchrony data obtained from the echocardiogram.

The dyssynchrony data will not be available to the treating physicians and will not be used to direct the LV lead location.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic CMP based on evidence of prior MI by history, coronary angiography/revascularization or imaging
* AHA ACC or ESC EHRA Guideline-based indication (Class I or II) for CRT and NYHA class II-IV heart failure
* ECG wide QRS and :

QRS > 120 msec in NYHA III- IV

OR

CLBBB or QRS > 150 in NYHA =II

* Sinus rhythm predominant rhythm (PAF not an exclusion)
* All must be candidates for De novo CRT-D implantation with LV lead via transvenous approach or patients previously implanted with pacemaker or ICD with <20% pacing over the last three months who are undergoing CRT-D upgrade.
* Patient provides informed consent, tolerate a pectoral implant, agree to comply with the protocol, and maintain scheduled follow-up visits.

Exclusion Criteria:

* Permanent or persistent atrial fibrillation
* Advanced renal disease (Cr >=2.5 mg/dL)
* Advanced comorbidities with life expectancy of <1 year
* Patients on waiting list for heart transplantation
* Requiring intravenous amines (continuous or or intermittent amine drip therapy)
* Severe chronic pulmonary disease (simulating heart failure)
* Severe (untreated) organic mitral valve disease
* Poorly treated hypertension
* History of myocardial infarction < 3 months; unstable angina < 1m, CABG <3 months; PCI <3 months
* Mechanical TC valve
* Previously implanted CRT system
* Poorly visualized cardiac chamber dimensions in an echocardiogram performed prior to enrollment - please help us define
* Pregnancy or child-bearing potential in the absence of accepted forms of birth control
* Concurrent enrollment in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Demonstrating Percent reduction in left ventricular end systolic (LVESV) at 6 months compared with baseline values. | within 12 month from enrollment.
  To show that in patients with ischemic cardiomyopathy, implantation of a CRT LV lead guided by radial strain imaging results in a significantly greater echocardiographic and clinical response to cardiac resynchronization therapy compared with conventional implantation techniques.

SECONDARY OUTCOMES:
Clinical Improvement | Within 12 month from enrollment
  A combined clinical event rate - change in NYHA, hospitalization for heart failure, death
Echocardiographic improvement | Within 12 month from enrollment
  >15% improvement in LVESV, >10% improvement in LVEDV, 5% absolute improvement of LVEF
Improvement in wellbeing | Within 12 month from enrollment
  10 point improvement in Minnesota Living with Heart Failure Questionnaire (MLWHF), 10% improvement of 6 minute walk test(6MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Goldenberg, Prof., Study Director — The Israeli Society for the Prevention of Heart Attacks; Michael Glikson, Prof., Principal Investigator — Sheba Medical Center; Paul Friedman, Prof., Principal Investigator — Mayo Clinic
Locations (9):
- Mayo Clinic, Rochester, Minnesota, United States
- Israel (8):
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Shaare Zedek, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Sorasky Medical Center, Tel Aviv

REFERENCES:
- [Background] Yu CM, Sanderson JE, Gorcsan J 3rd. Echocardiography, dyssynchrony, and the response to cardiac resynchronization therapy. Eur Heart J. 2010 Oct;31(19):2326-37. doi: 10.1093/eurheartj/ehq263. Epub 2010 Aug 13. PMID 20709721
- [Background] Miyazaki C, Redfield MM, Powell BD, Lin GM, Herges RM, Hodge DO, Olson LJ, Hayes DL, Espinosa RE, Rea RF, Bruce CJ, Nelson SM, Miller FA, Oh JK. Dyssynchrony indices to predict response to cardiac resynchronization therapy: a comprehensive prospective single-center study. Circ Heart Fail. 2010 Sep;3(5):565-73. doi: 10.1161/CIRCHEARTFAILURE.108.848085. Epub 2010 Jul 20. PMID 20647479
- [Background] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170
- [Background] Delgado V, van Bommel RJ, Bertini M, Borleffs CJ, Marsan NA, Arnold CT, Nucifora G, van de Veire NR, Ypenburg C, Boersma E, Holman ER, Schalij MJ, Bax JJ. Relative merits of left ventricular dyssynchrony, left ventricular lead position, and myocardial scar to predict long-term survival of ischemic heart failure patients undergoing cardiac resynchronization therapy. Circulation. 2011 Jan 4;123(1):70-8. doi: 10.1161/CIRCULATIONAHA.110.945345. Epub 2010 Dec 20. PMID 21173353
- [Background] Becker M, Hoffmann R, Kuhl HP, Grawe H, Katoh M, Kramann R, Bucker A, Hanrath P, Heussen N. Analysis of myocardial deformation based on ultrasonic pixel tracking to determine transmurality in chronic myocardial infarction. Eur Heart J. 2006 Nov;27(21):2560-6. doi: 10.1093/eurheartj/ehl288. Epub 2006 Oct 11. PMID 17035253
- [Background] Delgado V, Ypenburg C, van Bommel RJ, Tops LF, Mollema SA, Marsan NA, Bleeker GB, Schalij MJ, Bax JJ. Assessment of left ventricular dyssynchrony by speckle tracking strain imaging comparison between longitudinal, circumferential, and radial strain in cardiac resynchronization therapy. J Am Coll Cardiol. 2008 May 20;51(20):1944-52. doi: 10.1016/j.jacc.2008.02.040. PMID 18482662
- [Background] Tanaka H, Nesser HJ, Buck T, Oyenuga O, Janosi RA, Winter S, Saba S, Gorcsan J 3rd. Dyssynchrony by speckle-tracking echocardiography and response to cardiac resynchronization therapy: results of the Speckle Tracking and Resynchronization (STAR) study. Eur Heart J. 2010 Jul;31(14):1690-700. doi: 10.1093/eurheartj/ehq213. Epub 2010 Jun 8. PMID 20530502
- [Background] Kirn B, Jansen A, Bracke F, van Gelder B, Arts T, Prinzen FW. Mechanical discoordination rather than dyssynchrony predicts reverse remodeling upon cardiac resynchronization. Am J Physiol Heart Circ Physiol. 2008 Aug;295(2):H640-6. doi: 10.1152/ajpheart.00106.2008. Epub 2008 May 30. PMID 18515652
- [Background] Wang CL, Wu CT, Yeh YH, Wu LS, Chang CJ, Ho WJ, Hsu LA, Luqman N, Kuo CT. Recoordination rather than resynchronization predicts reverse remodeling after cardiac resynchronization therapy. J Am Soc Echocardiogr. 2010 Jun;23(6):611-20. doi: 10.1016/j.echo.2010.03.012. Epub 2010 Apr 24. PMID 20418055
- [Background] Wang CL, Powell BD, Redfield MM, Miyazaki C, Fine NM, Olson LJ, Cha YM, Espinosa RE, Hayes DL, Hodge DO, Lin G, Friedman PA, Oh JK. Left ventricular discoordination index measured by speckle tracking strain rate imaging predicts reverse remodelling and survival after cardiac resynchronization therapy. Eur J Heart Fail. 2012 May;14(5):517-25. doi: 10.1093/eurjhf/hfs025. Epub 2012 Mar 12. PMID 22411692
- [Background] Sung RK, Foster E. Assessment of systolic dyssynchrony for cardiac resynchronization therapy is not clinically useful. Circulation. 2011 Feb 15;123(6):656-62. doi: 10.1161/CIRCULATIONAHA.110.954420. No abstract available. PMID 21321181
- [Background] Kindermann M, Frohlig G, Doerr T, Schieffer H. Optimizing the AV delay in DDD pacemaker patients with high degree AV block: mitral valve Doppler versus impedance cardiography. Pacing Clin Electrophysiol. 1997 Oct;20(10 Pt 1):2453-62. doi: 10.1111/j.1540-8159.1997.tb06085.x. PMID 9358487